CLINICAL TRIAL: NCT04041505
Title: Feeding Infants in Nova Scotia: an Exploratory Analysis of Responsive Feeding With Mother's Milk
Brief Title: Responsive Feeding of Infants With Expressed Milk
Acronym: REFINE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Interim analysis (n=40 24-hr sessions) yielded biologically implausible data. We do not deem this novel, at-home, participant-led method prudent. Study will continue with only secondary objectives; primary objective (RCT) terminated.
Sponsor: Mount Saint Vincent University (Other)
Collaborators: University of Prince Edward Island (Other); Queen's University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: MSVUREB2018-155
Record Dates: First submitted 2019-07-04; First posted 2019-08-01 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-05

CONDITIONS: Human Milk; Breastfeeding; Feeding Behavior
Keywords: responsive feeding; expressing/pumping human milk
MeSH Terms: conditions — Breast Feeding; Feeding Behavior

STUDY DESIGN:
Intervention Model Description: This is a modified, randomized cross-over study. The 'intervention' in this study is simply feeding infants using one of two modalities that are already familiar to the mother and infant: feeding mother's milk from the breast and from a bottle.
  At each timepoint (6 weeks, 4 months, 6 months) infants will: be randomized using a balanced design (to control for order effect) to consume human milk from a bottle or from the breast for 24 hours; will then undergo a wash-out period in which they will be fed human milk as they usually would for 24 hours; then will complete the second 'treatment' (bottle or breast) for 24 hours. Due to the nature of the intervention, this study will not be blinded.
  We aim to recruit 62 mother-infant pairs (= 124 participants in total).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breastfeeding (Active Comparator): Infant consumes mother's milk directly from the breast.
  Interventions: Behavioral: (feeding modality)
- Bottle-feeding (Experimental): Infant consumes mother's expressed milk from a bottle.
  Interventions: Behavioral: (feeding modality)

INTERVENTIONS:
Behavioral: (feeding modality) — The intervention is a change in feeding modality: in both arms, infant's will consume mother's milk. The difference in arms is the modality in which human milk is consumed: either directly from the breast, or from a bottle.

SUMMARY:
Nova Scotia has among the lowest breastfeeding rates in Canada, with less than one quarter of infants receiving Health Canada's recommended 6 months of exclusive breastfeeding. Compared with feeding formula, breastfeeding has been linked with a number of health advantages, including fewer infections, higher IQ, and a lowered risk of obesity later in life.

How infants consume human milk is changing. Pumping milk has grown in popularity in recent years because some mothers may feel stigmatized breastfeeding, especially in public, but also because it allows other caregivers to help with feeding. Although pumped human milk is considered equal to breastfeeding, there is very little research in this area, especially around responsive feeding and later health outcomes. Since pumped milk is fed from a bottle, the health benefits may be lost (for instance, this may impact a baby's ability to understand if s/he is hungry or full).

The primary aim of this study is to determine if the volume of human milk an infant consumes differs if they consume milk from a bottle versus the breast. The investigators will conduct a cross-over trial in which 62 mother-infant pairs will be randomized to feed at the breast or from a bottle for 24 hours, have a 24 hour wash-out period, and then 'cross-over' to another 24 hour session with the opposite 'treatment.' The volume of milk consumed at each feed within the 24 hour window (via indirect weighing, or weighing the baby before and after eating) will be recorded to determine if there are differences in milk consumption. Mother-infant pairs will complete this 3-day study three times, at 6 weeks, 4 months, and 6 months.

Information from this study will help to better understand current infant feeding practices in Nova Scotia, and the potential role this plays in future health outcomes. Evidence from this study may help to identify means of improving feeding practices and promoting human milk as the main food for Nova Scotian infants, setting them on a path for the best start in life.

DETAILED DESCRIPTION:
See attached full protocol document for full details.

ELIGIBILITY:
Inclusion criteria: Mother-infant dyads are eligible to participate if:

* mother is aged 19 years or older,
* dyads currently live in the Halifax Regional Municipality in Nova Scotia,
* mother has no chronic diseases,
* the baby is a healthy singleton baby who is younger than 6 weeks of age, and is fed mother's milk directly from the breast and from a bottle,
* mother plans to exclusively feed their baby mother's own milk up to 6 months,
* mother has/had an older child whom they successfully fed mother's own milk for a minimum of 6 months,
* mother is willing to participate in three 3-day study sessions and monthly measurement sessions, and
* mother provides informed consent for herself and her infant to participate.

Exclusion criteria: Mother-infant dyads are ineligible to participate if:

* the baby was born preterm (earlier than 37 weeks gestation),
* the baby was born outside the healthy weight range of 2,500 - 4,000 g (5lb 8oz to 8lb 13oz),
* the baby has a developmental delay diagnosed before the time of enrolment,
* the baby is currently receiving any medical treatment except for vitamin D supplementation (no more than 400 IU/day),
* the mother sought prescription medical treatment for lactation (e.g. domperidone, antibiotics, prescription nipple ointment), or
* the mother plans to move in the 6 months after starting the study.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-08-15 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Volume of milk consumption | 24 hours
  To assess if the volume of human milk consumed by infants differs by feeding modality (bottle feeding human milk versus breastfeeding), assessed as overall milk volume consumed over 24 hours, measured by indirect weighs at each feed during a 24-hour period.

SECONDARY OUTCOMES:
Infant growth | Between 6 weeks and 6 months
  To determine whether change in infant anthropometric measurements (length in cm, weight in kg, head circumference in cm) and growth rates (weight-for-age [WAZ], length-for-age [LAZ], weight-for-length [WLZ], BMI-for-age z-scores [BAZ]; all computed as z-scores) differ by self-reported usual feeding modality among infants exclusively consuming human milk.
Responsive feeding behaviors | Between 6 weeks and 6 months
  To objectively assess responsiveness of infant feeding practices, both at the breast and during bottle-feeding of human milk, by video-recording feeding sessions in participant's homes.

OTHER OUTCOMES:
Feeding environment | Between 6 weeks and 6 months
  To gain a better understanding of current infant feeding practices, including responsive feeding, among caregivers in the Halifax Regional Municipality, contextualize why women are pumping, and gain insight around how human milk is handled, stored, and prepared through open-ended one-on-one interviews with mothers.

CONTACTS AND LOCATIONS:
Overall Officials: Kyly C Whitfield, PhD, Principal Investigator — Mount Saint Vincent University
Locations (1):
- MAMA Lab, Mount Saint Vincent University, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2019-09-27): https://cdn.clinicaltrials.gov/large-docs/05/NCT04041505/Prot_ICF_001.pdf